CLINICAL TRIAL: NCT06615674
Title: The Effect of Dapagliflozin on the Apoptosis Levels of Patients With Acute Myocardial Infarction - DAPOPTOSIS-MI (a Randomized Controlled Trial)
Brief Title: Effect of Dapagliflozin Administration on the Apoptosis Levels of Patients With Acute Myocardial Infarction
Acronym: DAPOPTOSIS-MI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yoga Yudhistira (Other)
Responsible Party: Sponsor-Investigator, Yoga Yudhistira, Principal Investigator, Universitas Sebelas Maret
Organization: Universitas Sebelas Maret (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S5121020014865
Record Dates: First submitted 2024-09-21; First posted 2024-09-26 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction (AMI); STEMI - ST Elevation Myocardial Infarction (MI); NSTEMI - Non-ST Segment Elevation Myocardial Infarction (MI)
Keywords: AMI; STEMI; NSTEMI; Dapagliflozin; Apoptosis; Caspase-3; Myocardial Work
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Spinocerebellar Ataxias | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial and Double Blind (Researcher &amp;amp;amp;amp;amp; Patients)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Experimental): The intervention group will have dapagliflozin 10mg once a day every morning besides standard treatment of Acute Coronary Syndrome for 14 days before further evaluation
  Interventions: Drug: Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia
- Control (Experimental): The first group is the Dapagliflozin group, which will get Dapagliflozin 10mg once a day every morning for 14 days. And the second group will have placebo for 14 days.
  Interventions: Drug: Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia

INTERVENTIONS:
Drug: Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia — The first group is the Dapagliflozin group, which will get Dapagliflozin 10mg once a day every morning for 14 days. And the second group will have placebo for 14 days.

SUMMARY:
The currently known Sodium-Glucose Transporter 2 (SGLT-2) inhibitors are recognized not only for their effects on improving intravascular glucose levels but also for their cardioprotective effects, including improvements in endothelial dysfunction, inhibition of platelet activation, reduction in autophagy processes, oxidative stress, and inflammation, as well as inhibition of the Na+/H+ exchanger pathway, which potentially reduces cell damage and death resulting from ischemia and reperfusion processes. Research on the benefits of SGLT-2 inhibitors in pre-clinical studies with myocardial infarction has shown a significant reduction in myocardial apoptosis, indicated by reduced levels of caspase-3 and the apoptosis index. Additionally, there was an increase in ketone bodies and myocardial ATP, reduced levels of inflammatory cytokines, free radicals, and infarct area, as well as improvements in left ventricular ejection fraction. However, large-scale studies in humans have thus far been limited to investigating the effects of SGLT-2 inhibitors on mortality, rehospitalization rates due to heart failure, cardiometabolic factors, and improvements in remodeling parameters in myocardial infarction patients, with the use of empagliflozin or dapagliflozin. Based on literature reviews, there have been no studies to date that directly demonstrate the effects of dapagliflozin on apoptosis (caspase-3 levels) in myocardial infarction patients.

DETAILED DESCRIPTION:
The study is a randomized controlled trial, single-center study in Acute Myocardial Infarction (AMI) patients held in Moewardi General Hospital, Central Java, Indonesia. The investigator divided 40 patients with AMI into two groups, the first is the Dapagliflozin group, which will get 10mg of Dapagliflozin once a day every morning and the second group will have a placebo once a day every morning also for 14 days. Each patient will be checked for Caspase-3 level from blood serum as primary outcome and Global Work (GW) echocardiographic parameters such as GWI, GCW, GWW, and GWE as secondary outcome at admission and 14 days after intervention. The study was approved by the hospital ethics committee. The clinical parameters above will then be analyzed. To determine the mean difference between unpaired groups (treatment and control), an independent T-test is used if the distribution is normal (if not, the Mann-Whitney test is used). Normality testing is performed using the Shapiro-Wilk test, considering the sample size is less than 50.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Acute Myocardial Infarction (STEMI or NSTEMI) according to the Fourth Universal Definition of Myocardial Infarction from the European Society of Cardiology, American College of Cardiology, American Heart Association, and World Heart Federation.
2. Aged 18-75 years
3. Willing to participate in the study and sign informed consent.

Exclusion Criteria:

1. Patients with cardiogenic shock (SBP ≤ 80 mmHg, cold extremities, urine output <0.5 ml/kg/hr) <24 hours before randomization
2. Patients with ketoacidosis (arterial pH <7.30, serum bicarbonate <18 mEq/l, positive ketonuria)
3. Patients with impaired renal function with an estimated glomerular filtration rate (eGFR) <20 ml/min or requiring dialysis
4. Patients with a history of chronic heart failure before the onset of Acute Myocardial Infarction
5. Patients scheduled for coronary artery bypass surgery
6. Patients with type 1 diabetes mellitus
7. Patients with severe valvular disease
8. Patients with sepsis
9. Patients with symptomatic acute urinary tract infection
10. Pregnant patients
11. Patients with severe aortic stenosis or LVOT obstruction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-21 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Change in Biomolecular Parameters | 14 days
  Change in Caspase-3 (ng/L) level in blood serum patients

SECONDARY OUTCOMES:
Change in Echocardiographic Parameters | 14 days
  Change in Global Work Index (GWI) (mmHg%), Global Constructive Work (GCW) (mmHg%), Global Wasted Work (GWW) (mmHg%), Global Work Efficiency (GWE) (%) parameter from patients

CONTACTS AND LOCATIONS:
Overall Officials: Yoga Yudhistira MD, Principal Investigator — Dr. Moewardi General Hospital, Jebres, Surakarta, Central of Java, 57126; Ahmad Yasa MD, Study Director — Dr. Moewardi General Hospital, Jebres, Surakarta, Central of Java, 57126
Locations (1):
- Dr. Moewardi General Hospital, Jebres, Surakarta, Central of Java, 57126, Surakarta, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
This study was conducted as part of the final project for the cardiovascular residency program, there was no sponsorship during this study therefore the IPD cannot be shared

REFERENCES:
- [Background] James S, Erlinge D, Storey RF, McGuire DK, de Belder M, Eriksson N, Andersen K, Austin D, Arefalk G, Carrick D, Hofmann R, Hoole SP, Jones DA, Lee K, Tygesen H, Johansson PA, Langkilde AM, Ridderstrale W, Parvaresh Rizi E, Deanfield J, Oldgren J. Dapagliflozin in Myocardial Infarction without Diabetes or Heart Failure. NEJM Evid. 2024 Feb;3(2):EVIDoa2300286. doi: 10.1056/EVIDoa2300286. Epub 2023 Nov 11. PMID 38320489
- [Background] Hernandez AF, Udell JA, Jones WS, Anker SD, Petrie MC, Harrington J, Mattheus M, Seide S, Zwiener I, Amir O, Bahit MC, Bauersachs J, Bayes-Genis A, Chen Y, Chopra VK, A Figtree G, Ge J, G Goodman S, Gotcheva N, Goto S, Gasior T, Jamal W, Januzzi JL, Jeong MH, Lopatin Y, Lopes RD, Merkely B, Parikh PB, Parkhomenko A, Ponikowski P, Rossello X, Schou M, Simic D, Steg PG, Szachniewicz J, van der Meer P, Vinereanu D, Zieroth S, Brueckmann M, Sumin M, Bhatt DL, Butler J. Effect of Empagliflozin on Heart Failure Outcomes After Acute Myocardial Infarction: Insights From the EMPACT-MI Trial. Circulation. 2024 May 21;149(21):1627-1638. doi: 10.1161/CIRCULATIONAHA.124.069217. Epub 2024 Apr 6. PMID 38581389
- [Background] Tanajak P, Sa-Nguanmoo P, Sivasinprasasn S, Thummasorn S, Siri-Angkul N, Chattipakorn SC, Chattipakorn N. Cardioprotection of dapagliflozin and vildagliptin in rats with cardiac ischemia-reperfusion injury. J Endocrinol. 2018 Feb;236(2):69-84. doi: 10.1530/JOE-17-0457. Epub 2017 Nov 15. PMID 29142025
- [Background] Jin W, Wang L, Zhu T, Ma Y, Yu C, Zhang F. Usefulness of echocardiographic myocardial work in evaluating the microvascular perfusion in STEMI patients after revascularization. BMC Cardiovasc Disord. 2022 May 13;22(1):218. doi: 10.1186/s12872-022-02648-z. PMID 35562649
- [Background] Chen S, Coronel R, Hollmann MW, Weber NC, Zuurbier CJ. Direct cardiac effects of SGLT2 inhibitors. Cardiovasc Diabetol. 2022 Mar 18;21(1):45. doi: 10.1186/s12933-022-01480-1. PMID 35303888
- [Background] McIlwain DR, Berger T, Mak TW. Caspase functions in cell death and disease. Cold Spring Harb Perspect Biol. 2015 Apr 1;7(4):a026716. doi: 10.1101/cshperspect.a026716. No abstract available. PMID 25833847
- [Background] Teringova E, Tousek P. Apoptosis in ischemic heart disease. J Transl Med. 2017 May 1;15(1):87. doi: 10.1186/s12967-017-1191-y. PMID 28460644